CLINICAL TRIAL: NCT05730036
Title: An Open-label, Randomized, Phase 3 Study of Linvoseltamab (REGN5458; Anti- BCMA x Anti-CD3 Bispecific Antibody) Versus the Combination of Elotuzumab, Pomalidomide, and Dexamethasone (EPd), in Patients With Relapsed/Refractory Multiple Myeloma (LINKER-MM3)
Brief Title: A Trial to Learn How Well Linvoseltamab Works Compared to the Combination of Elotuzumab, Pomalidomide and Dexamethasone for Adult Participants With Relapsed/Refractory Multiple Myeloma
Acronym: LINKER-MM3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R5458-ONC-2245; 2022-501396-62-00 (Registry Identifier: CTIS Number)
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-10

CONDITIONS: Relapsed Refractory Multiple Myeloma (RRMM)
Keywords: BCMA X CD3 Bispecific Monoclonal Antibody; CD38 antibody; Proteasome inhibitor; Lenalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab; pomalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Linvoseltamab (Experimental): Randomization 1:1
  Interventions: Drug: Linvoseltamab
- Elotuzumab/Pomalidomide/Dexamethasone (EPd) (Active Comparator): Randomization 1:1
  Interventions: Drug: Elotuzumab; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Linvoseltamab — REGN5458 will be administered by intravenous (IV) infusion
  Other Names: REGN5458; Lynozyfic™
  Arms: Linvoseltamab
Drug: Elotuzumab — Elotuzumab will be administered by IV infusion
  Other Names: Empliciti
  Arms: Elotuzumab/Pomalidomide/Dexamethasone (EPd)
Drug: Pomalidomide — Pomalidomide capsules will be administered by mouth (PO)
  Other Names: Pomalyst
  Arms: Elotuzumab/Pomalidomide/Dexamethasone (EPd)
Drug: Dexamethasone — Dexamethasone tablets/capsules will be administered PO and/or by IV infusion
  Other Names: Decadron
  Arms: Elotuzumab/Pomalidomide/Dexamethasone (EPd)

SUMMARY:
This study is researching an experimental drug called linvoseltamab, also called REGN5458.

Linvoseltamab has previously been studied by itself (without other cancer drugs) in participants who had advanced multiple myeloma that returned and needed to be treated again after many other therapies had failed. These participants were no longer benefiting from standard medications and had no good treatment options. In that study, some participants who were treated with linvoseltamab had improvement of their myeloma (shrinkage of their tumors), including some participants who had complete responses (that is, the treatment got rid of all evidence of myeloma in their bodies).

This study is focused on participants who have multiple myeloma that has returned or needs to be treated again after one to four prior treatments and have standard cancer treatment options available to them. The aim of this study is to see how safe and effective linvoseltamab is compared to a combination of three cancer drugs: elotuzumab, pomalidomide and dexamethasone, (called EPd) in participants who have returned after having received prior treatment that included lenalidomide, a proteosome inhibitor, and (for participants in some countries) a cluster of differentiation 38 (CD38) antibody. Half of the participants in this study will get linvoseltamab, and the other half will get EPd.

This study is looking at several other research questions, including:

* How long participants benefit from receiving linvoseltamab compared with EPd
* How many participants treated with linvoseltamab or EPd have improvement of their multiple myeloma and by how much
* What side effects happen from taking linvoseltamab compared to EPd
* How long participants live while receiving treatment or after treatment with linvoseltamab compared to EPd
* If there is any improvement in pain after treatment with linvoseltamab compared to EPd

ELIGIBILITY:
Key Inclusion Criteria:

1. Age 18 years or older (or legal adult age in the country) at the time of the screening visit.
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤1. Patients with ECOG 2 solely due to local symptoms of myeloma (eg. pain) may be allowed after discussion with the Medical Monitor.
3. Received at least 1 and no more than 4 prior lines of anti-neoplastic MM therapies, including lenalidomide and a proteasome inhibitor and demonstrated disease progression on or after the last therapy as defined by the 2016 IMWG criteria. Participants who have received only 1 line of prior line of antimyeloma therapy must be lenalidomide refractory, as described in the protocol.

   Note: Participants in Israel also must have previously received a CD38 antibody. Participants in the EU and the UK must have previously received 2 to 4 prior lines of therapy, including a CD38 antibody.
4. Patients must have measurable disease for response assessment as per the 2016 IMWG response assessment criteria, as described in the protocol
5. Adequate hematologic function and hepatic function within 7 days of randomization, as well as adequate renal and cardiac function and corrected calcium
6. Life expectancy of at least 6 months

Key Exclusion Criteria:

1. Diagnosis of plasma cell leukemia, amyloidosis, Waldenström macroglobulinemia, or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
2. Prior treatment with elotuzumab and/or pomalidomide
3. Participants with known MM brain lesions or meningeal involvement
4. Treatment with any systemic anti-cancer therapy within 5 half-lives or within 28 days before first administration of study drug, whichever is shorter
5. History of allogeneic stem cell transplantation within 6 months, or autologous stem cell transplantation within 12 weeks of the start of study treatment. Participants who have received an allogeneic transplant must be off all immunosuppressive medications for 6 weeks without signs of graft-versus-host disease. Steroids at doses equivalent to suppletion doses may be acceptable.
6. Prior treatment with B-cell maturation antigen (BCMA) directed immunotherapies Note: BCMA antibody-drug conjugates are allowed.
7. History of progressive multifocal leukoencephalopathy (PML), known or suspected PML, or history of a neurocognitive condition or central nervous system (CNS) movement disorder (Parkinson's disease or Parkinsonism).
8. Any infection requiring hospitalization or treatment with IV anti-infectives within 2 weeks of first administration of study drug
9. Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV); or another uncontrolled infection, as defined in the protocol 10 Cardiac ejection fraction <40%.

NOTE: Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2033-04-19 (Estimated); Study Completion 2033-04-19 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) per International Myeloma Working Group (IMWG) response criteria determined by Independent Review Committee (IRC) in CD38 antibody exposed participants | Up to approximatively 5 years

SECONDARY OUTCOMES:
PFS per IMWG response criteria determined by IRC in all participants | Up to approximatively 5 years
Objective Response (OR) of Complete Response (CR) or better per IMWG response criteria as determined by IRC in CD38 antibody exposed participants | Up to approximatively 5 years
OR of CR or better per IMWG response criteria as determined by IRC in all participants | Up to approximatively 5 years
Overall Survival (OS) in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
OS in all participants | Up to approximatively 5 years
Incidence of minimal residual disease (MRD) negative status in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
Incidence of MRD negative status in all participants | Up to approximatively 5 years
Mean change in the worst pain score measured by Brief Pain Inventory-Short Form (BPI-SF) Item 3 in participants previously exposed to CD38 antibodies | Baseline to week 12
  The BPI-SF is a validated, self-administered questionnaire designed to measure a participant's perceived level of pain. The BPI-SF Item 3 uses a numeric rating scale to assess pain severity and pain interference in the past 24 hours. The numeric rating scale ranges from 0 (no pain) to 10 (worst imaginable pain), where higher scores indicate greater intensity of pain.
Mean change in the worst pain score measured by BPI-SF Item 3 in all participants | Baseline to week 12
  The BPI-SF is a validated, self-administered questionnaire designed to measure a participant's perceived level of pain. The BPI-SF Item 3 uses a numeric rating scale to assess pain severity and pain interference in the past 24 hours. The numeric rating scale ranges from 0 (no pain) to 10 (worst imaginable pain), where higher scores indicate greater intensity of pain.
Incidence of treatment emergent adverse events (TEAEs) in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
Incidence TEAEs in all participants | Up to approximatively 5 years
Severity of TEAEs in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
Severity of TEAEs in all participants | Up to approximatively 5 years
Incidence of adverse events of special interest (AESI) in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
Incidence of AESI in all participants | Up to approximatively 5 years
Severity of AESI in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
Severity AESI in all participants | Up to approximatively 5 years
Incidence of Serious Adverse Events (SAE) in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
Incidence of SAE in all participants | Up to approximatively 5 years
Severity of SAE in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
Severity of SAE in all participants | Up to approximatively 5 years
PFS per IMWG response criteria as determined by the investigator in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
PFS per IMWG response criteria as determined by the investigator in all participants | Up to approximatively 5 years
OR of Partial Response (PR) or better per IMWG response criteria as determined by the IRC in CD38 antibody exposed participants | Up to approximatively 5 years
OR of PR or better per IMWG response criteria as determined by the IRC in all participants | Up to approximatively 5 years
OR of Very Good Partial Response (VGPR) or better per IMWG response criteria as determined by IRC in CD38 antibody exposed participants | Up to approximatively 5 years
OR of VGPR or better per IMWG response criteria as determined by IRC in all participants | Up to approximatively 5 years
OR of PR or better per IMWG response criteria as determined by the investigator in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
OR of PR or better per IMWG response criteria as determined by the investigator in all participants | Up to approximatively 5 years
OR of VGPR or better per IMWG response criteria as determined by the investigator in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
OR of VGPR or better per IMWG response criteria as determined by the investigator in all participants | Up to approximatively 5 years
OR of CR or better per IMWG response criteria as determined by the investigator in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
OR of CR or better per IMWG response criteria as determined by the investigator in all participants | Up to approximatively 5 years
Duration of Response (DoR) as per IMWG response criteria as determined by the investigator in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
DoR as per IMWG response criteria as determined by the investigator in all participants | Up to approximatively 5 years
DoR as per IMWG response criteria as determined by the IRC in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
DoR as per IMWG response criteria as determined by the IRC in all participants | Up to approximatively 5 years
Duration of MRD negative status in the bone marrow in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
Duration of MRD negative status in the bone marrow in all participants | Up to approximatively 5 years
Time from randomization to objective response (≥PR) as per IMWG response criteria as determined by the investigator in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
Time from randomization to objective response (≥PR) as per IMWG response criteria as determined by the investigator in all participants | Up to approximatively 5 years
Time from randomization to objective response (≥PR) as per IMWG response criteria as determined by the IRC in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
Time from randomization to objective response (≥PR) as per IMWG response criteria as determined by the IRC in all participants | Up to approximatively 5 years
Concentration of linvoseltamab in the serum over time in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
Concentration of linvoseltamab in the serum over time in all participants | Up to approximatively 5 years
Incidence of antidrug antibodies (ADAs) in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
Incidence of ADAs in all participants | Up to approximatively 5 years
Titer of ADAs in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
Titer of ADAs in all participants | Up to approximatively 5 years
Incidence of neutralizing antibodies (Nabs) to linvoseltamab over time in participants previously exposed to CD38 antibodies | Up to approximatively 5 years
Incidence of Nabs to linvoseltamab over time in all participants | Up to approximatively 5 years
Proportion of Pain Responders in participants previously exposed to CD38 antibodies | At week 12
  Defined by at least a 2-point reduction from baseline in the BPI-SF Item 3 without an increase in analgesic use using the modified Analgesic Quantification Algorithm (AQA).
Proportion of Pain Responders in all participants | At week 12
  Defined by at least a 2-point reduction from baseline in the BPI-SF Item 3 without an increase in analgesic use using the modified Analgesic Quantification Algorithm (AQA).
Change in patient-reported global health status/quality of life (QoL), per European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) in participants previously exposed to CD38 antibodies | Baseline to week 12
  The EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including global health status/quality of life, functional Scales (physical, role, emotional, cognitive, and social), symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participants rate items on a 4-point scale, with 1 as "not at all" and 4 as "very much."
Change in patient-reported QoL, per EORTC QLQ-C30 in all participants | Baseline to week 12
  The EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including global health status/quality of life, functional Scales (physical, role, emotional, cognitive, and social), symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participants rate items on a 4-point scale, with 1 as "not at all" and 4 as "very much."
Change in patient reported disease symptoms per EORTC Quality of Life Questionnaire-Multiple Myeloma (MM) module 20 [QLQ-MY20]) in participants previously exposed to CD38 antibodies | Baseline to week 12
  The EORTC QLQ-MY20 is a self -administered instrument to assess QoL in persons with MM. This 20-item questionnaire measures the following domains: symptom scales, including disease symptoms (6 items) and symptoms related to side effects of treatment (10 items); function scale and future perspective (3 items); and body image (1 item). A high score represents a high level of symptoms or problems.
Change in patient reported disease symptoms per EORTC QLQ-MY20 in all participants | Baseline to week 12
  The EORTC QLQ-MY20 is a self -administered instrument to assess QoL in persons with MM. This 20-item questionnaire measures the following domains: symptom scales, including disease symptoms (6 items) and symptoms related to side effects of treatment (10 items); function scale and future perspective (3 items); and body image (1 item). A high score represents a high level of symptoms or problems.
Patient-Reported Outcomes in Patient Global Impression of Symptom Severity (PGIS) in participants previously exposed to CD38 antibodies | Baseline to week 12
  The PGIS is a single 1-item questionnaire designed to assess participant's overall impression of disease severity at a given point in time by using a 4-point Likert scale that ranges from (1) = "none (no symptoms)" to (4) = "severe".
  The global anchor, PGIS will be used for interpretation of EORTC QLQ-C30, EORTC QLQ-MY20, and BPI-SF.
Patient-Reported Outcomes in PGIS in all participants | Baseline to week 12
  The PGIS is a single 1-item questionnaire designed to assess participant's overall impression of disease severity at a given point in time by using a 4-point Likert scale that ranges from (1) = "none (no symptoms)" to (4) = "severe".
  The global anchor, PGIS will be used for interpretation of EORTC QLQ-C30, EORTC QLQ-MY20, and BPI-SF.
Patient-Reported Outcomes in Patient Global Impression of Change (PGIC) in participants previously exposed to CD38 antibodies | Baseline to week 12
  The PGIC is a single-item questionnaire designed to assess the participant's overall sense of whether there has been a change since starting treatment as rated on a 5-point Likert scale anchored by (1) "much better" to (5) "much worse", with (4) = "no change".
  The global anchor, PGIC will be used for interpretation of EORTC QLQ-C30, EORTC QLQ-MY20, and BPI-SF.
Patient-Reported Outcomes in PGIC in all participants | Baseline to week 12
  The PGIC is a single-item questionnaire designed to assess the participant's overall sense of whether there has been a change since starting treatment as rated on a 5-point Likert scale anchored by (1) "much better" to (5) "much worse", with (4) = "no change".
  The global anchor, PGIC will be used for interpretation of EORTC QLQ-C30, EORTC QLQ-MY20, and BPI-SF.
Change in patient-reported general health status per EuroQoL-5 Dimension-5 Level Scale [EQ-5D-5L]) in participants previously exposed to CD38 antibodies | Baseline to week 12
  The EQ-5D-5L consists of EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Change in patient-reported general health status per EQ-5D-5L in all participants | Baseline to week 12
  The EQ-5D-5L consists of EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (158):
- United States (10):
  - University of California Los Angeles (UCLA), Los Angeles, California
  - University of Florida Division of Sponsored Programs, Gainesville, Florida
  - University of Kentucky, Markey Cancer Center Clinical Research Organization, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Stony Brook University, Stony Brook, New York
  - Levine Cancer Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Kaiser Permanente Northwest, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas
  - University of Washington, Seattle, Washington
- Australia (11):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Icon Cancer Centre - Wesley, Auchenflower, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Launceston General Hospital, Launceston, Tasmania
  - St Vincent's Hospital, Fitzroy, Victoria
  - University Hospital Geelong, Geelong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - One Clinical Research at Hollywood Private Hospital, Nedlands, Western Australia
- Belgium (4):
  - Clinique Universitaire de Mont Godinne, Yvoir, Namur
  - AZ Delta Algemeen Ziekenhuis Delta, Roeselare, West-Vlaanderen
  - Ziekenhuis Netwerk Antwerpen Stuivenberg, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
- Brazil (11):
  - IDOR - Sao Rafael Salvador Bahia, Salvador, Estado de Bahia
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Associacao Dr Bartholomeu Tacchini, Bento Gonçalves, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Centro Gaucho Integrado, Porto Alegre, Rio Grande do Sul
  - Animi Unidade de Tratamento Oncologico, Lages, Santa Catarina
  - Instituto Americas de Ensino e Pesquisa, Rio de Janeiro
  - A Beneficencia Portuguesa de Sao Paulo, Oncology House, São Paulo
  - Instituto DOr de Pesquisa e Ensino, São Paulo
  - AC Camargo Cancer Center, São Paulo
  - Clinica Medica Sao Germano, São Paulo
- Canada (3):
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Cancer Center, Toronto, Ontario
- Chile (6):
  - Hospital Clinico Universidad de Los Andes, Santiago, Las Condes
  - Centro de Investigaciones Clinicas Vina del Mar, Viña del Mar, Región de Valparaíso
  - Clinica Alemana de Santiago, Santiago, Santiago Metropolitan
  - Fundacion Arturo Lopez Perez, Santiago, Santiago Metropolitan
  - Clinica UC San Carlos de Apoquindo, Santiago, Santiago Metropolitan
  - Centro Oncologia de Precision Universidad Mayor, Santiago, Santiago Metropolitan
- France (8):
  - Centre Leon Berard (CLB) - Centre de Recherche en Cancerologie Lyon-Est (CRCL), Lyon, Auvergne-Rhone
  - Centre Francois Magendie, Pessac, Gironde
  - Centre Hospitalier Universitaire de Lille, Lille, Hauts-de-France
  - Hopital Saint Louis, APHP, Paris
  - Saint Antoine Hospital, Paris
  - Institut Curie, Saint-Cloud
  - Hopital Necker, Paris, Île-de-France Region
  - Gustave Roussy, Villejuif, Île-de-France Region
- Germany (4):
  - Medical Clinic II, Tübingen, Baden-Wurttemberg
  - Universitat zu Lubeck Neuromuskulares Zentrum, Lübeck, Ratzeburger
  - University Hospital Hamburg Eppendorf, Hamburg
  - University Hospital Leipzig - Hematology and Cellular Therapy, Leipzig
- Israel (6):
  - Rambam Health Care Campus, Haifa, North
  - Lady Davis Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - The Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (13):
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Istituto Romagnolo per lo Studio Dei Tumori Dino Amadori, Meldola, Forli-Cesena
  - Ospedale Policlinico San Martino IRCCS, Genoa, Genova
  - Azienda Ospedaliera Nazionale SS - Antonio e Biagio e Cesare Arrigo, Alessandria, Piedmont
  - A.O.U. Citta della Salute e della Scienza di Torino, Turin, Piedmont
  - IRCCS Fondazione Piemontese Oncologica Candiolo, Candiolo, Torino
  - AOU Ospedali Riuniti di Ancona, Ancona
  - Policlinico S. Orsola- Malpighi, Bologna
  - Azienda Ospedaliero Universitaria Policlinico "G. Rodolico - San Marco", Catania
  - Universita degli Studi di Pavia - Fondazione IRCCS Policlini, Pavia
  - Ospedale Santa Maria delle Croci, Ravenna
  - AUSL IRCCS OF Reggio Emilia - Clinical Study Location -, Reggio Emilia
  - Ospedale di Circolo e Fondazione Macchi Varese, Varese
- Japan (18):
  - Aichi Medial University Hospital, Nagakute, Aichi-ken
  - Chiba Cancer Center, Chiba, Chiba
  - Kameda General Hospital, Kamogawa, Chiba
  - Kurume University Hospital, Kurume, Fukuoka
  - Ogaki Municipal Hospital, Ōgaki, Gifu
  - Gunma University Hospital, Maebashi, Gunma
  - NHO Shibukawa Medical Center, Shibukawa, Gunma
  - Sapporo Hokuyu Hospital, Sapporo, Hokkaido
  - Iwate Medical University Hospital, Yahaba, Iwate
  - National Hospital Organization Kumamoto Medical Center, Kumamoto, Kumamoto
  - National Hospital Organization Okayama Medical Center, Kita-ku, Okayama-ken
  - Osaka University Hospital, Suita-shi, Osaka
  - Saitama Medical University Hospital, Iruma-gun, Saitama
  - Tokushima Prefectural Central Hospital, Tokushima, Tokushima
  - Japanese Red Cross Medical Center, Shibuya-ku, Tokyo
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
  - Fukushima Medical University, Fukushima
  - National Hospital Organization Sendai Medical Center, Sendai
- Netherlands (2):
  - Radboudumc, Nijmegen, Gelderland
  - Albert Schweitzer Hospital, Dordrecht, South Holland
- Poland (5):
  - University Clinical Center / Medical University of Gdansk, Gdansk, Pomeranian Voivodeship
  - Szpital Uniwersytecki Nr2 Bydgoszcz, Bydgoszcz
  - Pratia Onkologia Katowice, Katowice
  - Centrum Innowacyjnych Terapii Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - Wielospecjalistyczne Centrum Onkologii i Traumatologii, Lodz, Łódź Voivodeship
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
- South Korea (10):
  - Gachon University Gil Hospital, Incheon, Gyeonggi-do
  - Jeonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Inje University Busan Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Asan Medical Center, Seoul
  - Seoul St Marys Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
- Spain (27):
  - Hospital Clinico Universitario Santiago de Compostela, Santiago de Compostela, A Coruna
  - Hospital Universitario Araba, Vitoria-Gasteiz, Alava
  - Hospital Universitari Son Espases, Palma, Balearic Islands
  - Hospital Universitari Son Llatzer, Palma Mallorca, Balearic Islands
  - Institut Catala d'Oncologia, Badalona, Barcelona
  - Hospital Universitari Mutua Terrassa, Terrassa, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Complejo Asistencial Universitario de Leon, León, Castille and León
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Clinica Universidad de Navarra - Pamplona, Pamplona, Navarre
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - University Hospital of Cabuenes, Gijón, Principality of Asturias
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Universitary Hospital La Princesa, Madrid, Salamanca
  - Hospital General Universitario Doctor Balmis Alicante, Alicante, Valencia
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Sant Pau, Barcelona
  - Catalan Institute of Oncology (ICO) Hospitalet, Barcelona
  - Instituto Catalan Oncologia, Girona
  - Clinica Universidad de Navarra - Madrid, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Clinico Lozano Blesa, Zaragoza
- Taiwan (10):
  - Chang Gung Memorial Hospital - Linkou Branch, Taoyuan District, Hunan Province
  - Changhua Christian Hospital, Changhua
  - Hualien Tzu Chi Hospital, Hualien City
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Wanfang Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- United Kingdom (8):
  - Addenbrooke's Hospital, Cambridge, Cambrigeshire
  - Western General Hospital, Edinburgh, Scotland
  - Queen Elizabeth Hospital Birmingham, Birmingham, West Midlands
  - Barts Health NHS Trust, London
  - Guy's & St Thomas' NHS Foundation Trust, London
  - Royal Marsden Hospital, London
  - Hammersmith Hospital, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: Study Information Website — https://linkerclinicalstudies.com/en-us